CLINICAL TRIAL: NCT03451929
Title: Kidney Function and Markers of Inflamation in Relation to Mortality, Cardiovascular Events and Kidney Function Impaired: Cohort Study in General Adult Population
Brief Title: Kidney Function and Cardiovascular Events: Cohort Study in General Population
Acronym: EPIRCE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: María Pilar Gayoso Diz (Other)
Responsible Party: Sponsor-Investigator, María Pilar Gayoso Diz, Family Medicine, PhD, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Other Study IDs: EPIRCE2; PI13/02031 (Other Grant/Funding Number: IS Carlos III)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Diseases; Progression; Cardiovascular Morbidity
Keywords: primary healthcare; cohort
MeSH Terms: conditions — Renal Insufficiency, Chronic; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine samples with DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective multicenter follow-up study of 10 years. Cohort established between 2005-2007 with stratified random sample of general population older than 20 years (Census 2001), N= 2746 subjects.

DETAILED DESCRIPTION:
The aim of this study is to analyse the evolution of kidney function (KF) in the general Spanish population and its impact in terms of quality of life, survival and prognosis for relevant clinical events: mortality, major vascular events and end stage renal disease (ESRD), over a period of 10 years. This is in line with the research priorities highlighted by Kidney Disease: Improving Global Outcomes (KDIGO) 2012.

The study is a prospective multi-centre 10 year follow-up study. Cohort established in Phase I of the EPIRCE study conducted in 2005-2007; stratified random sample of the general population over age 20 (2001 Census), with 2746 subjects studied with complete baseline characterization: socio-demographic variables, lifestyle factors, vascular risk, morbidity, and RF. Cox proportional hazard additive predictors will be used to study the predictive value of renal function models. All models will be adjusted for socio-demographic factors and lifestyle. IDI and NRI will be used to determine whether the addition of KF improves the predictive ability of the existing scores. Decision curve analysis will be used to indicate different KF cut-off points take cost and benefit into account in the decision to treat or not treat.

This project addresses the predictive capacity of glomerular filtration and albuminuria on mortality and vascular events after a 10-year follow-up in the general population, with an analysis of potential improvement in predicting vascular mortality and/or major vascular events by incorporating renal function into existing scales. It also establishes associated serum DNA samples to a well phenotyped cohort for subsequent studies of gene expression and inflammatory markers on CKD. These results will therefore provide insight into the natural evolution of CKD and associated vascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Subjects studied in Phase I of the EPIRCE study. Give their informed consent to participate in this phase of EPIRCE 2 study.

Exclusion Criteria:

* Exclusion criteria: subjects that cannot be located or who refuse to give their consent to participate in this monitoring phase will be excluded.

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A random sample, stratified by age and sex, of the over 20 population, representative of the general adult Spanish population. The sample population was the 2001 Census (National Statistical Institute of Spain, INE).
  Sample size: 2746 subjects studied in Phase I of the EPIRCE study are included. This sample size allows for a 1.17% accuracy rate for the estimate of a proportion (prevalence) in a maximum dispersion variable (p = q = 0.5) with a 95% confidence interval.
Sampling Method: Probability Sample
Enrollment: 2746 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Impaired renal function | 2005-2018, up to 10 years
  50% reduction in the glomerular filtration rate with respect to the baseline
mortality | 2005-2018, up to 10 years
  mortality due to cardiovascular problems or any others
ACS | 2005-2018, up to 10 years
  acute coronary syndrome
stroke | 2005-2018, up to 10 years
  ischemic, due to lack of blood flow, and hemorrhagic, due to bleeding.

SECONDARY OUTCOMES:
health related quality of life | 2014-2018
  SF-12
depression or anxiety | 2014-2018
  Hospital Anxiety Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Gayoso-Diz, PhD, Principal Investigator — National Health Service of Spain

IPD SHARING:
Plan to Share IPD: No